CLINICAL TRIAL: NCT06859190
Title: Analysis of the Efficacy of Auricular Pressure Beans Combined with Electroacupuncture and Estazolam for the Treatment of Insomnia Induced by Cancer
Brief Title: Efficacy of Auricular Pressure Beans with Electroacupuncture and Estazolam Treating Insomnia Caused by Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qinghai Red Cross Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-03
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Insomnia
Keywords: cancer; auricular pressure beans; electroacupuncture; insomnia; estazolam
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Estazolam; Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ONS group) (Experimental): Patients will receive estazolam with auricular pressure points and electroacupuncture treatment.
  Interventions:In the experimental group, estazolam (oral estazolam 1-2 mg daily at bedtime) was combined with auricular pressure point therapy and electroacupuncture over an 8-week period.
  Interventions: Drug: estazolam 1-2 mg; Procedure: Auricular pressure bean combined with electroacupuncture
- Arm II (NS group) (Active Comparator): Patients will follow the standard estazolam treatment program(oral estazolam 1-2 mg daily at bedtime for 8 weeks).
  Interventions: Drug: estazolam 1-2 mg

INTERVENTIONS:
Drug: estazolam 1-2 mg — oral estazolam 1-2 mg daily at bedtime for 8 weeks.
Procedure: Auricular pressure bean combined with electroacupuncture — Electroacupuncture treatment will be performed on seven acupoints, including Baihui (GV20), Shenting (GV24), Yintang (GV29), Anmian (EX-HN22), Shenmen (HT7), Neiguan (PC6), and Sanyinjiao (SP6). Each session lasts for 30 minutes and is conducted twice a week.In addition, auricular point seed-pressing therapy will be applied to bilateral auricular points related to insomnia (Shenmen, Heart, and Sympathetic). Each auricular point will be pressed for 1 minute, three times a day. The total treatment course is eight weeks.
  Arms: Arm I (ONS group)

SUMMARY:
The core objectives of this study are to assess the short-term and long-term efficacy of auricular acupoint pressure beans combined with electroacupuncture and estazolam in the treatment of cancer-caused insomnia. The study aims to accurately compare the differences between this combination therapy and standard Western medicine in improving sleep quality and effectively alleviating anxiety and depression. Additionally, it will meticulously observe the safety of the combined treatment and record the occurrence and potential causative factors of any adverse reactions.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled, open-label clinical trial evaluating the efficacy of auricular pressure beans combined with electroacupuncture and estazolam in treating cancer-caused insomnia. A total of 60 patients will be enrolled and randomized into a control group and an experimental group, each consisting of 30 patients.Patients in the control group will follow the standard estazolam treatment program, with the drug dosage adjusted according to individual conditions to achieve the best therapeutic effect. In the experimental group, auricular pressure points and electroacupuncture will be skillfully integrated with estazolam treatment. The auricular pressure points will be carefully selected based on their relation to insomnia (e.g., Shenmen, heart, sympathetic) and will be replaced once or twice a week. Electroacupuncture will target key acupoints such as Baihui, Shenmen, and Sanyinjiao, with each session lasting 30 minutes and conducted twice a week.Data collection will involve the Insomnia Severity Index, Pittsburgh Sleep Quality Index (PSQI), Hamilton Anxiety Scale (HAMA), Hamilton Depression Rating Scale (HAMD), and other assessments through questionnaires and clinical evaluations at the end of the 0th, 4th, and 8th weeks of treatment, as well as during follow-up (12th, 16th, and 20th weeks). All adverse reactions occurring throughout the treatment process will be closely monitored and recorded, including both drug-related and non-drug-related adverse reactions. Professional statistical software will be used to analyze the data rigorously, comparing dynamic changes in various indicators between the experimental and control groups before and after treatment, thereby scientifically assessing the efficacy and safety of the combined treatment for cancer-related insomnia. This rigorous study design and comprehensive data analysis aim to provide new perspectives and evidence for treating cancer-related insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above.
2. The diagnosis of a malignant solid tumor was confirmed by pathological examination.
3. Clinically diagnosed cancer-caused insomnia with insomnia symptoms lasting more than 1 month, more than 3 or more times per week.
4. An Insomnia Severity Index (ISI) score of 8 or higher and meets the criteria for insomnia disorder as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition.
5. No medications related to the treatment of insomnia have been used in the last 1 month.
6. No serious dysfunction of the heart, liver, kidneys or other vital organs.
7. Patients volunteered to participate in this study and signed an informed consent form.

Exclusion Criteria:

1. Irregular sleep-wake cycles in jobs with shift demands or due to inconsistent work schedules.
2. Inadequately treated for another sleep disorder (e.g., sleep disorder disorders such as sleep apnea obstruction syndrome, restless leg syndrome, etc.).
3. Received acupuncture or auricular pressure bean therapy within the past 3 months.
4. Estimated life expectancy is ≥3 months.
5. Have a history of severe allergies, especially to the drugs or treatments used in this study.
6. History of severe mental illness with a current episode.
7. History of substance abuse or alcohol dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The Insomnia Severity Index(ISI) | Data will be collected at the end of the 0th, 4th, and 8th weeks of treatment and during follow-up (12th, 16th, and 20th weeks).
  The scale is a simple tool used for screening insomnia, consisting of 7 items designed to assess the nature and symptoms of sleep disturbances in the subjects.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index(PSQI) | Data will be collected at the end of the 0th, 4th, and 8th weeks of treatment and during follow-up (12th, 16th, and 20th weeks).
  The Pittsburgh Sleep Quality Index (PSQI) is used to assess the sleep quality of subjects over the past month . It consists of 9 self-rated items and 5 other-rated items, with a total of 18 items grouped into 7 factors. Each factor is scored on a scale of 0 to 3, and the cumulative scores of the factor components make up the total score of the Pittsburgh Sleep Quality Index. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Hamilton Anxiety Scale(HAMA) | Data will be collected at the end of the 0th, 4th, and 8th weeks of treatment and during follow-up (12th, 16th, and 20th weeks).
  The Hamilton Anxiety Scale (HAMA) includes 14 items and is one of the most widely used clinician-administered scales in psychiatry. It is primarily used to assess the severity of anxiety symptoms in patients with neuroses and other conditions.
Hamilton Depression Rating Scale(HAMD) | Data will be collected at the end of the 0th, 4th, and 8th weeks of treatment and during follow-up (12th, 16th, and 20th weeks).
  The scale includes 24 items and is primarily scored through the clinician's observation and questioning of the patient, aiming to provide a comprehensive assessment of various aspects of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- China, Qinghai,Qinghai Red Cross Hospital, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: Undecided